CLINICAL TRIAL: NCT03429465
Title: Training Resiliency in Youth (TRY) Study
Acronym: TRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Pat Arean, Professor, School of Medicine: Psychiatry And Behavioral Sciences, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00003107
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Attention Concentration Difficulty; Depression; Anxiety
Keywords: Digital Health Intervention; Executive Function; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EVO (Experimental): All children receive 4 weeks of EVO 5 days/week for 20 minutes per day in a stepped wedge design.
  Interventions: Other: EVO Cognitive Remediation Game

INTERVENTIONS:
Other: EVO Cognitive Remediation Game — EVO (formerly called Neuroracer) is a neuroscience-inspired plasticity trainings in the form of a video driving game that uses adaptive algorithms and dual-tasking paradigms to target the CCN. Work from our group (Project:EVO) recently showed that 4 weeks of EVO training is associated with increased neural recruitment in brain regions associated with CNN, superior improvement in cognitive control performance (i.e., working memory, sustained attention) when compared to an evidence-based psychotherapy (Problem-Solving Therapy), and improved depression outcomes similar to Problem-Solving Therapy among older adults (Areán, Hallgren, Jordan, Gazzaley, Atkins, Heagerty, & Anguera, 2016; Journal of Medical Internet Research).

SUMMARY:
The aim of the study is to determine whether a neuroscience-inspired cognitive remediation video game (EVO) that targets the cognitive control network (CCN) will improve executive functioning (EF) and resilience to psychiatric symptoms in typically developing 6th grade students, unselected for specific psychiatric symptoms. The primary goals are to 1) determine if EVO will result in improved EF and lower internalizing (e.g., mood, anxiety) and externalizing (e.g., attention deficit/hyperactivity disorder, AD/HD) psychiatric symptoms, 2) evaluate whether the benefit experienced by youth changes depending on their level of life stress (e.g., academic or social difficulties), 3) determine if EVO will promote resilience to stress. The investigators will measure EF, symptoms, and stress using self- and parent-report questionnaires. Other secondary outcomes include information on behavior in the classroom and academic performance (i.e., grades) that we will collect via school records. The investigators hypothesize that engagement with EVO 20-minutes per day, 5-days a week across 4-weeks will improve EF, lower psychiatric symptoms, improve academic/behavioral functioning at school, and decrease maladaptive responses to stress.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in 6th grade during the 2017-2018 school year at Lucille Umbarger Elementary School in the Burlington-Edison School District
* Physical ability to use a touchscreen iPad
* Cognitive ability to assent, complete questionnaires, and play EVO game
* English speaking child, English or Spanish speaking parent
* Child has legal parent/guardian (i.e., not a ward of the state)

Exclusion Criteria:

* The child is identified by parent or school as diagnosed with an intellectual disability
* The child is identified by parent or school as diagnosed with a physical disability (i.e., unable to use hands or fingers) that would preclude use of a touchscreen iPad and appropriate engagement with EVO
* The child is identified by parent or school as unlikely to engage for 20 minutes with EVO
* Child unable to read or understand English
* Parent unable to read or understand English/Spanish
* Child is in public (i.e., child welfare) custody

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-06-04 (Actual); Study Completion 2018-06-04 (Actual)

PRIMARY OUTCOMES:
Executive Function | Measured 5 times across 5 months
  Measuring Executive Function (e.g., attention, working memory) via parent-report of children's symptoms.
Behavioral Problems | Measured 5 times across 5 months
  Measuring difficulties with attention (i.e., attention deficit/hyperactivity disorder), oppositionality, and conduct at home and school as measured by parent-report on children's behavior.
Depression | Measured 5 times across 5 months
  depression symptoms measured with self- and parent- report
Anxiety | Measured 5 times across 5 months
  Measuring self- and parent-reported symptoms of anxiety.

SECONDARY OUTCOMES:
Emotion Regulation | Measured 5 times across 5 months
  Measuring self-reported cognitive aspects of emotion regulation (e.g., rumination, positive reappraisal).

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Arean, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States